CLINICAL TRIAL: NCT00860925
Title: PeriOperative ISchemic Evaluation-2 (POISE-2) Trial: A Pilot
Brief Title: PeriOperative ISchemic Evaluation-2 Pilot
Acronym: POISE2-pilot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Canadian Network and Centre for Trials Internationally (Unknown)
Responsible Party: Dr P.J. Devereaux, McMaster University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POISE-2 01 2009
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Cardiovascular Disease
Keywords: Randomized Controlled Trial; Blinded; Clonidine; acetyl-salicylic acid (ASA); Perioperative vascular complications; Noncardiac surgery
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- active clonidine and active ASA (Experimental)
  Interventions: Drug: active clonidine; Drug: active ASA
- active clonidine and ASA placebo (Experimental)
  Interventions: Drug: active clonidine; Drug: ASA Placebo
- Clonidine placebo and active ASA (Experimental)
  Interventions: Drug: active ASA; Drug: Clonidine Placebo
- Clonidine placebo and ASA placebo (Placebo Comparator)
  Interventions: Drug: Clonidine Placebo; Drug: ASA Placebo

INTERVENTIONS:
Drug: active clonidine — Prior to surgery (goal 2-4 hours) patients will ingest 1 tablet of clonidine (0.2 mg) and will have a transdermal clonidine patch (0.2 mg/day) applied. The patch will be removed at 72 hours after surgery.
  Other Names: CATAPRES, CATAPRES TTS
  Arms: active clonidine and ASA placebo; active clonidine and active ASA
Drug: active ASA — Prior to surgery (goal 2-4 hours) patients will ingest 2 ASA tablets (81 mg per tablet). After the first dose, patients will ingest 1 tablet daily for 7 or 30 days according to the stratum they are allocated to. Patients who are not able to take ASA orally will receive it rectally.
  Other Names: ENTROPHEN CHEWABLE
  Arms: Clonidine placebo and active ASA; active clonidine and active ASA
Drug: Clonidine Placebo — Prior to surgery (goal 2-4 hours) patients will take oral clonidine placebo and will have a transdermal placebo patch applied. The patch will be removed at 72 hours after surgery.
  Other Names: CATAPRES placebo and CATAPRES TTS placebo
  Arms: Clonidine placebo and ASA placebo; Clonidine placebo and active ASA
Drug: ASA Placebo — Prior to surgery (goal 2-4 hours) patients will ingest 2 ASA placebo tablets. After the first dose, patients will ingest 1 placebo tablet daily for 7 or 30 days according to the stratum they are allocated to. Patients who are not able to take placebo orally will receive it rectally.
  Other Names: ENTROPHEN CHEWABLE placebo
  Arms: Clonidine placebo and ASA placebo; active clonidine and ASA placebo

SUMMARY:
Major non-cardiac surgeries are common and major heart problems during or after such surgeries represent a large population health problem. Few treatments to prevent heart problems around the time of surgery have been tested.

There is encouraging data suggesting that low-doses of Acetyl-Salicylic Acid (ASA) and Clonidine, which are two medications, given individually for a short period before and after major surgeries may prevent major heart problems.

DETAILED DESCRIPTION:
The POISE-2 Pilot Trial will provide the essential remaining feasibility data that POISE-2 researchers require prior to conducting a large international study to test the effect of ASA and Clonidine in preventing major vascular complications during the first 30 days after surgery.

The POISE-2 Pilot Trial is a factorial design randomized control trial that will compare ASA to placebo and clonidine to placebo. Patients in the POISE-2 pilot trial will be randomly assigned to one of four groups: ASA and Clonidine together, ASA and Clonidine placebo, ASA placebo and Clonidine, or a ASA placebo and Clonidine placebo. Two to four hours prior to surgery, eligible patients are given ASA study drug and Clonidine study drug orally (162mg ASA or its placebo and 0.2mg Clonidine or its placebo) and a patch to apply (0.2mg/day Clonidine or its placebo). The patch will remain in place for 72 hours after surgery. After the surgery, patients ingest one tablet a day (81mg ASA or its placebo) for 7 days if patient was were taking ASA chronically prior to surgery or for 30 days if they were not chronically taking ASA prior to surgery. Troponin measurements will be collected between 6 to 12 hours after the operation and on the 1st, 2nd, and 3rd days after surgery. If blood tests reveal an elevation in the troponin measurement an electrocardiogram (ECG) will be undertaken immediately.

Research personnel will follow patients until 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing noncardiac surgery who fulfill the following criteria:

* age ≥ 45 years
* expected to require at least an overnight hospital admission after noncardiac surgery, and fulfill any 1 of the following criteria:

  * history of coronary artery disease
  * peripheral vascular disease
  * stroke
  * undergoing major vascular surgery (i.e., vascular surgery except arteriovenous shunt, vein stripping procedures, and carotid endarterectomies)
  * OR any 3 of 9 risk criteria:

    1. undergoing major surgery [i.e., intraperitoneal, intrathoracic, or orthopedic surgery]
    2. history of congestive heart failure
    3. transient ischemic attack
    4. diabetes and currently taking an oral hypoglycemic agent or insulin
    5. age = or > than 70 years
    6. hypertension
    7. serum creatinine > 175 µmol/L
    8. history of smoking within 2 years of surgery, or
    9. undergoing emergent/urgent surgery

Exclusion Criteria:

* Patients has taken ASA < or = to 72 hours before scheduled surgery
* history of ASA or clonidine hypersensitivity or allergy
* systolic blood pressure < 105 mm Hg
* heart rate < 55 beats per minute
* second or third degree heart block without a pacemaker
* patient has active peptic ulcer disease
* Patient has had a bare metal stent in the six weeks prior to randomization
* Patient has had a drug eluting stent in the year prior to randomization
* Patient is currently taking an alpha-2 agonist, alpha methyldopa, reserpine, clopidogrel, or ticlopidine
* Patient undergoing intracranial surgery, carotid endarterectomy, or retinal surgery
* Surgeon unwilling to have patient participate in a participate in a perioperative clonidine/ASA trial
* Prior enrolment in the POISE-2 pilot trial
* Unable to obtain or refusal to consent prior to surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting 90 patients in 6 months | 6 months

SECONDARY OUTCOMES:
Feasibility of administering pre-operative ASA and clonidine | 6 months
Preliminary estimate of major bleeding and clinically significant hypotension | 30 days
Preliminary estimate of the composite of vascular death and non-fatal myocardial infarction. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: P. J. Devereaux, MD FRCP PHD, Principal Investigator — McMaster University
Locations (4):
- Canada (3):
  - Walter C MacKenzie Health Sciences, Edmonton, Alberta
  - Hamilton Health Sciences, Hamilton, Ontario
  - St Joseph's Health Sciences, Hamilton, Ontario
- Prince of Wales Hospital, Hong Kong, China